CLINICAL TRIAL: NCT01699048
Title: Prospective, Single-center, Randomized Trial, Intended to Compare Three Revascularization Strategies in Patients With Multi-vessel Coronary Artery Disease
Brief Title: The Comparative Effectiveness of Hybrid Revascularization (MIDCAB Then PCI) With DES Versus Multivessel DES PCI or CABG
Acronym: HREVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr. Vladimir Ganyukov, Hybrid minimally invasive and Interventional coronary revascularization in patients with Multi-vessel coronary artery disease versus complete Endovascular Revascularisation or coronary Artery bypass graft (treatment strategies)., Russian Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREVS
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases
Keywords: multivessel PCI,MIDCAB,CABG; Hybrid coronary revascularization
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hybrid group (Other): Hybrid approach (Minimally invasive off-pump revascularization of the left anterior descending artery (LAD) with the left internal mammary artery (LIMA) bypass followed by consecutive percutaneous coronary intervention (PCI) in the rest of the arteries with drug eluting stents (DES) (Hybrid group, n=50)
  Interventions: Procedure: Hybrid (MIDCAB+PCI)
- PCI (Other): Multi-vessel PCI with DES (MV-PCI group, n=50)
  Interventions: Procedure: PCI
- CABG (Other): Coronary artery bypass graft (CABG) treatment (CABG group, n=50)
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: Hybrid (MIDCAB+PCI) — Hybrid approach (Minimally invasive of-pump revascularization of the left anterior descending artery (LAD) via left internal mammary artery (LIMA) bypass with consecutive percutaneous coronary intervention (PCI) in the rest arteries with drug eluting stents (DES). The revascularization will be performed in two stages within a 3-days interval
  Other Names: MIDCAB
  Arms: Hybrid group
Procedure: PCI — Multi-vessel PCI with DES
  Arms: PCI
Procedure: CABG — Coronary artery bypass graft (CABG) treatment
  Arms: CABG

SUMMARY:
Minimally invasive revascularization of the left anterior descending artery followed by stent implantation versus percutaneous coronary intervention or coronary artery bypass in patients with multi-vessel coronary disease

DETAILED DESCRIPTION:
Prospective, single-center, randomized trial, intended to compare three revascularization strategies in patients with multi-vessel coronary artery disease:

1. Hybrid approach (Minimally invasive off-pump revascularization of the left anterior descending artery (LAD) with left internal mammary artery (LIMA) bypass followed by consecutive percutaneous coronary intervention (PCI) in the rest of the arteries with drug eluting stents (DES) (Hybrid group, n=50)
2. Multi-vessel PCI with DES (MV-PCI group, n=50)
3. Coronary artery bypass graft (CABG) treatment (CABG group, n=50)

PCI in Hybrid and MV-PCI group will be performed with the same 2nd generation clinically proven DES (Xience V, Xience Prime).

Study objective Compare three different revascularization strategies in patients with multi-vessel coronary disease

The endpoints:

The primary endpoints:

I. % ischemic myocardium on a 12-month follow-up scan with single photon emission computed tomography (SPECT);

The secondary endpoints:

I. Major adverse cardiac and cerebral events (MACCE), including (1) death, (2) non-fatal myocardial infarction (non-fatal MI), transitory ischemic attack (TIA) or stroke within 30 days, 12 months and 5-year follow-up; II. Target vessel/graft failure (for any of the target vessels in a given patient - stented or grafted) = a composite of cardiac death, MI attributable to the target vessel, or clinically-driven [ie, not angio-driven] Target Vessel Revascularization (TVR); III. Restenosis = angiographically-detected target lesion stenosis >50% [diameter stenosis] or graft stenosis >50%; IV. Procedural success: The treatment will be considered successful when a revascularisation in the absence of complications during the index hospitalization has been achieved; V. Procedural and post-procedural hemorrhagic complications [ Time Frame: up to discharge from the hospital ]; VI. Recovery time [ Time Frame: up to discharge from the hospital ];

ELIGIBILITY:
Inclusion Criteria:

1. Multi-vessel coronary artery disease with ≥ 70% and <96% artery stenosis (according to QCA)
2. I-IV CCS functional class of angina
3. Asymptomatic patients with stress-test documented ischemia.
4. Patients at 1 month after acute myocardial infarction
5. Ability to perform either of revascularization methods (Hybrid, MVD-PCI, CABG).
6. Consensus on the treatment strategy between the members of the working group, including cardiologist, cardiac surgeon and interventional specialist.
7. Patients must have signed an informed consent.

Exclusion Criteria:

1. Pregnancy.
2. Acute coronary syndrome.
3. Previous CABG.
4. Previous stent thrombosis.
5. Severe comorbidity with high procedural risk for either of the studied strategies.
6. Severe peripheral artery disease.
7. Other serious diseases limiting life expectancy (e.g. oncology)
8. Inability for long-term follow-up.
9. Participation in other clinical trials.
10. Inability to take dual antithrombotic therapy.

Angiographic exclusion criteria

1. Critical stenosis (>95%) in RCA,LAD, CX or Intermediate artery, feasible for revascularization.
2. Stenosis of left main ≥ 50%.
3. Coronary artery occlusion of the major vessel.
4. Single vessel disease.
5. Need for emergency revascularization (ACS).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-12-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-09-16 (Actual)

PRIMARY OUTCOMES:
Residual ischemia | 6 - to 18-month follow-up
  ≥5% residual ischemia by single photon emission computed tomography (SPECT)

SECONDARY OUTCOMES:
MACCE | up to 5 years
  Major adverse cardiac and cerebral events (MACCE), including death,a composite of major cardiac and cerebrovascular events, i.e. the first occurrence of any of the following events:
  Death from any cause From cardiovascular causes From noncardiovascular causes Stroke or transitory ischemic attack (TIA) MI Hospitalization for repeat revascularization procedure, target (vessel) revascularization by means of PCI or CABG.
Procedural success | up to discharge from the hospital
  Procedural success: The treatment will be considered successful when a complete hybrid revascularisation in the absence of complications during the index hospitalization has been achieved.
Procedural and post-procedural blood loss and number of transfusions | up to discharge from the hospital
  dynamics of hemoglobin at admission and discharge, the number of blood transfusions (in units), classification of bleeding BARC
Recovery time | up to discharge from the hospital
  Time Frame: from the end of the intervention up to discharge from the hospital. Total duration of hospital admission
Target vessel/graft failure | 6- to 18-month follow-up
  (for any of the target vessels in a given patient - stented or grafted) = a composite of cardiac death, MI attributable to the target vessel, or clinically-driven [ie, not angio-driven] Target Vessel Revascularization (TVR);
Restenosis | 6- to 18-month follow-up
  angiographically-detected target lesion stenosis >50% [diameter stenosis] or graft stenosis >50%;

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Complex Issues of Cardiovascular Diseases, Kemerovo, Kemerovo Oblast, Russia

REFERENCES:
- [Derived] Ganyukov VI, Kochergin NA, Shilov AA, Tarasov RS, Skupien J, Kozyrin KA, Barbarash OL, Musialek P. Randomized Clinical Trial of Surgical Versus Percutaneous Versus Hybrid Multivessel Coronary Revascularization: 3 Years' Follow-Up. JACC Cardiovasc Interv. 2021 May 24;14(10):1163-1165. doi: 10.1016/j.jcin.2021.02.037. No abstract available. PMID 34016423
- [Derived] Ganyukov V, Kochergin N, Shilov A, Tarasov R, Skupien J, Szot W, Kokov A, Popov V, Kozyrin K, Barbarash O, Barbarash L, Musialek P. Randomized Clinical Trial of Surgical vs. Percutaneous vs. Hybrid Revascularization in Multivessel Coronary Artery Disease: Residual Myocardial Ischemia and Clinical Outcomes at One Year-Hybrid coronary REvascularization Versus Stenting or Surgery (HREVS). J Interv Cardiol. 2020 Jan 3;2020:5458064. doi: 10.1155/2020/5458064. eCollection 2020. PMID 31969796